CLINICAL TRIAL: NCT03738956
Title: Safety and Efficacy of Tofacitinib in the Treatment of NSAID Refractory Axial Spondyloarthritis:A Clinical Trial
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Globe Pharmaceuticals Limited (Other)
Collaborators: Globe pharmaceuticals Ltd, Dhaka, Bangladesh (Unknown)
Responsible Party: Principal Investigator, Dr.Md.Asadul Islam, Resident, Globe Pharmaceuticals Limited
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BSMMU/2017/9442
Record Dates: First submitted 2018-11-08; First posted 2018-11-13 (Actual); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Axial Spondyloarthritis
Keywords: Axial spondyloarthritis
MeSH Terms: conditions — Axial Spondyloarthritis | interventions — tofacitinib

STUDY DESIGN:
Intervention Model Description: Eligible patients will be given tofacitinib 5 mg BD ,at the end of 1st and 3rd months they will be assessed for safety and efficacy.At 3rd months if any patient wll not responds then they will be given tofacitinib 10 mg BD,at the end of 6th month they will be assessed for safety and efficacy.If any adverse events occur they will be treated accordingly.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open label clinical trial (Experimental): NSAID refractory axial spondyloarthritis patients who are eligible after considering inclusion and exclusion crietria will be put on 5 mg tofacitinib BD ,at the end of 1st and 3rd month they will be assessed for safety and efficacy.Those who will not respond will be put on 10 mg tofacitinib BD.All patients will be assessed at the end of 6th month.If any adverse event occur they will be treated accordingly.
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: Tofacitinib — The study subjects fulfilling the inclusion criteria will receive tofacitinib 5mg BD.
  All the patients in the study group will go through disease history, clinical examination and baseline investigations. Baseline charachteristics and variables will be recorded at initiation of therapy, 4th, 12th and 24th week. Primary endpoint of efficacy will be assessed using ASAS 20 response at the end of 12 th wk. At the end of 12 th week, those patients will achieve primary endpoint will continue with the same dose and those patients who will not achieve primary endpoint will be put on tofacitinib10 mg BD. Those patients who will not respond to treatment at the end of 24 th wk will discontinue the therapy and put on alternative treatment.

SUMMARY:
Title Efficacy and Safety of Tofacitinib in the Treatment of NSAID-Refractory Axial Spondyloarthritis: A Clinical Trial

Background:

Axial spondyloarthritis (axSpA) is a chronic systemic inflammatory rheumatic disease affecting mainly sacroiliac joints and spine. There are limited options for treatment. Initial treatments are patient's education, regular physical exercise and nonsteroidal antiinflammatory drugs(NSAID). If the patients do not respond to at least two NSAIDs in full dosages for at least one month then it is called NSAID refractory axSpA. In these cases biologics like-tumor necrosis factor α blockers are the options for treatment. Tofacitinib is a new drug has been proven to be effective for treatment of rheumatoid arthritis , psoriasis , inflammatory bowel disease and supposed to be effective in spondyloarthritis. This study is aimed to assess the efficacy and safety of tofacitinib in NSAID refractory ax SpA with a view to find a safe, effective and affordable treatment modality.

Method:

This open label uncontrolled clinical trial with tofacitinib will be conducted in NSAID refractory axSpA (age >18 years) patients. Study participants will be enrolled after having informed written consent from the outpatient department of Rheumatology, Bangabandhu sheikh mujib medical university. Assessment of Spondyloarthritis International Society (ASAS) criteria will be followed for diagnosis of ax SpA. Patients failing a trial of 2 different NSAID each for at least 2 weeks with optimum dosage without response or with partial response and Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score of ≥4 (range, 0-10) or Ankylosing spondylitis disease activity score-C reactive protein(ASDAS-CRP)>2.1 will be considered as primary entry criteria for this study.

Baseline evaluation will include Bath AS Disease Activity Index (BASDAI), Functional Index (BASFI) , Ankylosing spondylitis disease activity score-C reactive protein(ASDASCRP) and Ankylosing spondylitis disease activity score-erythrocyte sedimentation rate(ASDAS-ESR).

Laboratory tests like CBC, ESR, CRP, SGPT, Serum creatinine and X-ray pelvis A/P view or X-ray both SI joints modified Ferguson veiw (to see both SI and hip joints ), HLA-B27(if needed), CXR P/A view and MT test or Interferon Gamma Release Assay(IGRA) will be done.

After considering inclusion and exclusion criteria eligible patients will be included for this study. All patients will be put on 5mg tofacitinib BD. NSAID and adjuvant analgesics will be used if needed. Follow up will be done at 4th, 12th and 24th week. Response to treatment will be evaluated by assessement of spondyloarthritis society (ASAS) response criteria. More than 20% improvements from baseline will consider as primary response at the end of 12th week. Those patients who will not achieve ASAS20 response at 12th week, will be given 10 mg tofacitinib BD. Efficacy will be assessed at the end of 24th week by ASAS20, ASAS50, ASAS70, ASDAS-ESR, ASDAS-CRP, BASDAI, Bath ankylosing spondylitis functional index(BASFI). Adverse effects will be assesed by history, Physical examinations and investigations.

The entire study subjects will be informed about the nature, purpose and implication of the study as well as whole spectrum of benefits and risk of the study. Ethical clearance will be taken from the IRB of BSMMU.

DETAILED DESCRIPTION:
INTRODUCTION Spondyloarthritis (SpA) is one of the most prevalent forms of chronic inflammatory arthritis. It affects approximately 0.01-2.5% in the World wide. Estimated prevalence of SpA in India is between 0.1 to 0.2% and prevalence in Bangladesh is about 1.2% .

Janus kinase (JAK) is a family of intracellular, nonreceptor tyrosine kinase that transduce cytokine-mediated signals via theJAK-signal transduction and activation of transcriptors( JAK-STAT) pathway. The JAK-STAT signaling pathway transmits information from extracellular chemical signals to the nucleus resulting in DNA transcription and expression of genes involved in immunity, proliferation, differentiation, apoptosis and oncogenesis .

Tofacitinib acts by inhibiting JAK-STAT pathway particularly JAK1 and/JAK3 of multilineage cells thereby inhibiting lymphocytes. It inhibits interleukin IL-17, IL-21, IL-23 and interferon IFN-γ productions by CD4 T cells acts on dendritic cells(DCs) and suppressed inflammatory cytokine productions and expression of costimulatory molecules, also supprressed T cell stimulatory capacity of DCs. These indicate that wide range of biological effects of tofacitinib that directly and indirectly affect cytokine pathway thereby modulate immunue response and reduce inflammations.

Axial SpA patients treated with tofacitinib experienced clinically meaningful reductions in axial MRI inflammations and thereby an increased clinical response rates. A 16-week, phase II, randomized trial on AS patients with tofacitinib showed 80.8 % patients achieved ASAS 20 response .

As the therapeutic options of NSAID refractory axial SpA are limited, we want to assess the efficacy of tofacitinib in refractory axial SpA. In our country there are no studies of tofacitinib on axial spondyloarthritis. In Bangladesh, tofacitinib is cheaper than anti TNF biologics so it will reduce the treatment cost.

Rationale of the Study There are limited options for treating NSAID refractory axial SpA. Therefore, choosing the appropriate therapeutic options, efficacy, long term safety, and tolerability should be considered. Recently, biological agents having anti tumor necrosis factor-α (TNF-α) activity are now considered as 1st line treatment for refractory axial SpA. But these drugs are costly difficult to afford by most of the people of our country and there is also increase risk of activation of the latent tuberculosis, other adverse effects like malignancies, hematological disorders and various infections are still a problem. n our country this drug is less costly affordable by many people and as it is available as tablet form so drug compliance will be better than biological drugs.

Research Hypothesis

Null hypothesis:

Tofacitinib is not effective in NSAID refractory axial SpA.

Alternative hypothesis:

Tofacitinib is effective in the treatment of NSAID refractory axial SpA. Tofacitinib is safe in the treatment of NSAID refractory axial SpA.

Objectives Primary Objective To assess the efficacy and safety of tofacitinib in the treatment of NSAID refractory axial SpA

Secondary Objectives To compare the efficacy and safety of 10 mg and 20 mg tofacitinib in the treatment of NSAID refractory axial SpA.

Methodology Study Design: Open label uncontrolled clinical trial. Place of Study Out-patient department of Rheumatology, Bangabandhu Sheikh Mujib Medical University (BSMMU), Dhaka.

Study Period:

One and half year after IRB clearance

Study population:

Adult patients with back pain >3 months and age of onset of pain at <45yrs of age, attending outpatient department of rheumatology , BSMMU, who fullfill the ASAS classification criteria for axSpA and refractory to NSAID will be considered for the study.

Sample size calculation Information needed:

1. P1=Outcome of one group
2. P2= Outcome of another group
3. Zα= Z -value at a definite level of significance
4. Zβ = Z -value at a definite power. Formula: n = n = sample size for each group Sample size calculation for this study:(van der Heijde D, 2017) P1= 81% (0.81) P2= 41%(0.41)

Zα=1.96 at 5% level of significance Zβ= 1.28 at 90% power (when β=0.1) n =2.475x10.497 =25.96

Sample Size: A total 30 subjects will be included considering around10% dropout.

Sampling: Consecutive

Study Procedure An open labeled prospective, uncontrolled study will be conducted in outpatient Department of Rheumatology, BSMMU for 18 months (May 2017 to August 2018). Total 30 patients with NSAID refractory axial SpA will be enrolled in the study. Informed written consent will be obtained from all participants.

The study subjects fulfilling the inclusion criteria will receive tofacitinib 5mg BD.

All the patients in the study group will go through disease history, clinical examination and baseline investigations. Baseline charachteristics and variables will be recorded at initiation of therapy, 4th, 12th and 24th week. Primary endpoint of efficacy will be assessed using ASAS 20 response at the end of 12 th wk. At the end of 12 th week, those patients will achieve primary endpoint will continue with the same dose and those patients who will not achieve primary endpoint will be put on tofacitinib10 mg BD. Those patients who will not respond to treatment at the end of 24 th wk will discontinue the therapy and put on alternative treatment. All the baseline variables will be recorded and statistical analysis will be done.

Patients who develop serious drug related adverse effect like life threatening infection with organ involvement or requiring hospital admission will be withdrawn from the the study.

Safety assessment:

Clinical and laboratory parameters will be monitor at 1st, 3rd and 6th month.

Patient follow-up schedule:

Follow up will be done at the end of 4th, 12th and 24th week. At every follow up detailed history, thorough physical examination and some investigations will be done to evaluate the adverse effects.

Laboratory Investigations:

CBC, ESR, and CRP, S. creatinine, S. ALT and urine RME will be done during follow up.

Criteria for discontinuing a study participant:

A participant will be excluded from the study under following circumstances .If any patient fails to come for follow-up routinely. If patients develop toxicity -Severe adverse drug reactions, Infections (TB) etc. If patients stop to take the drug by themselves .

Variables:

Demographic variables

1. Age
2. Gender
3. Education
4. Occupation
5. Monthly income
6. BMI Outcome variables Assessement of Spondyloarthritis International Society-20(ASAS-20) response Assessement of Spondyloarthritis International Society-50(ASAS-50) response Assessement of Spondyloarthritis International Society-70(ASAS-70) response Ankylosing Spondylitis Disease Activity Score-CRP(ASDAS-CRP) Ankylosing Spondylitis Disease Activity Score-ESR(ASDAS-ESR) Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Bath Ankylosing Spondylitis Functional Index(BASFI) Duration of morning stiffness Patient global assessment & Physician global assessment on NRS/VAS Statistical analysis The degrees of statistical significance between the intragroup values of the endpoints will be analyzed by paired t test if the observations are normally distributed, otherwise it will be compared with paired Wilcoxon signed rank test. Probabilities of associations will be assessed by calculating Spearman's rank correlation coefficient. P values will be regarded as significant if they will <0.05.

Quality assurance strategy This will be uncontrolled clinical trial. Extensive literature search was done. Direct supervision by guide and co-guides will be done. Investigator will be sufficiently trained. Patient will purchase the drugs from pharmacy execpt tofacitinib which will provide free of cost and all of these drugs will be checked by the investigator. Monthly pill count will be done to ensure drug adherence. Patients will be educated properly not to take other medications that interact with tofacitinib(Rifampicin,ketoconazole) during the whole study period .During his/her follow up visit every time it will be ensured that he/she is not taking any other medication except those suggested by us. To prevent loss of follow up, telephone number of patient and caregiver will be collected, permanent and present address will be noted meticulously. They will advise to come for a follow up visit monthly. If any patient will miss it then he/she will be contacted over telephone to know their where about. If they are not available by telephone then a letter will be send to their present and permanent address. If they failed to reply and if they live nearby then I myself or a volunteer will be send to his/ her resident. Review of the study status will be done every fortnightly by the investigator with Guide. 10% data will be checked randomly by the guide. It will be an unbiased study. After collection, all data will be checked for inadequacy, irrelevancy and inconsistency. Irrelevant and inconsistent data will be discarded.

ELIGIBILITY:
Inclusion Criteria:

* The subjects will be considered if they fulfill the following criteria

  1. Subjects greater than 18 years of age
  2. Patients fulfilling the ASAS classification criteria for axial SpA including both non radiographic axial spondyloarthritis (nr-Ax SpA) and ankylosing spondylitis(AS)
  3. Patients with axSpA underwent a trial of at least 2 course of NSAIDs with optimum doses for at least 1 month without response or with partial response
  4. Patients with BASDAI ≥4 or ASDAS-CRP>2.1

Exclusion Criteria:

* The subjects will be excluded if they have any of the

  1. Systemic infections requiring hospital admission during the last 6 months
  2. Active infections and/or a history of chronic or recurrent serious infective diseases, opportunistic infections
  3. Hemoglobin (Hb) < 9 g/dl
  4. White blood cell count < 4000, Neutrophil count < 1000, Platelet count < 100000/mm3
  5. Live vaccines within 3 months prior to the first dose
  6. Serum creatinine > upper limit of normal reference range
  7. GFR less than 50 mL/min
  8. Alanine aminotransaminase (ALT) more than 2 times of ULN
  9. Pregnant or breast feeding females of child-bearing potential not using highly effective contraception
  10. Evidence or history of malignancy, with the exception of adequately treated or excised non-metastatic basal or squamous cell cancer of the skin or cervical carcinoma in situ
  11. New York Heart Association Class III and IV congestive heart failure
  12. Any lymphoproliferative disorder, history of lymphoma, leukemia, or signs and symptoms suggestive of current lymphatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-12-30 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of spondyloarthritis international society 20 response(ASAS 20) | At the end of 3rd month
  ASAS 20:It is a composite measurement which means improvement of ≥ 20% in 3 of the following 4 domains without 20% worsening in the remaining domain
  Four domains
  1. Bath ankylosing spondylitis functional index(BASFI)-The 10 items index of daily functional activities completed on a numerical rating scale (NRS) 0-10. The higher the BASFI score, the more severe the limitation of function due to AxSpA
  2. Morning stiffness
  3. Patient global assessment
  4. Pain

SECONDARY OUTCOMES:
Ankylosing Spondylitis Disease Activity Score- C reactive protein(ASDASCRP) | At the end of 6 month
  ASDAS-CRP: 0.121×total back pain+0.110×patient global+0.073×peripheral pain/swelling+0.058×duration of morning stiffness+0.579×Ln(CRP+1).
Ankylosing Spondylitis Disease Activity Score-Erythrocyte sedimentation rate(ASDASESR) | At the end of 6th month
  ASDAS-ESR: 0.113×patient global+0.293xESR----√+0.086×peripheral pain/swelling+0.069×duration of morning stiffness+0.079×total back pain.

CONTACTS AND LOCATIONS:
Overall Officials: Asadul Islam, MBBS, Principal Investigator — Globe Pharmaceuticals Limited
Locations (1):
- Bangabandhu sheikh mujib medical university, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Boonen A, van der Heijde D, Landewe R, Guillemin F, Rutten-van Molken M, Dougados M, Mielants H, de Vlam K, van der Tempel H, Boesen S, Spoorenberg A, Schouten H, van der Linden S. Direct costs of ankylosing spondylitis and its determinants: an analysis among three European countries. Ann Rheum Dis. 2003 Aug;62(8):732-40. doi: 10.1136/ard.62.8.732. PMID 12860728
- [Background] Anderson JJ, Baron G, van der Heijde D, Felson DT, Dougados M. Ankylosing spondylitis assessment group preliminary definition of short-term improvement in ankylosing spondylitis. Arthritis Rheum. 2001 Aug;44(8):1876-86. doi: 10.1002/1529-0131(200108)44:83.0.CO;2-F. PMID 11508441
- [Background] Sykes WS, Lawrence RC. Helium in Anaesthesia. Br Med J. 1938 Aug 27;2(4051):448-9. doi: 10.1136/bmj.2.4051.448. No abstract available. PMID 20781696
- [Background] Braun J, Pham T, Sieper J, Davis J, van der Linden S, Dougados M, van der Heijde D; ASAS Working Group. International ASAS consensus statement for the use of anti-tumour necrosis factor agents in patients with ankylosing spondylitis. Ann Rheum Dis. 2003 Sep;62(9):817-24. doi: 10.1136/ard.62.9.817. PMID 12922952
- [Background] Braun J, Inman R. Clinical significance of inflammatory back pain for diagnosis and screening of patients with axial spondyloarthritis. Ann Rheum Dis. 2010 Jul;69(7):1264-8. doi: 10.1136/ard.2010.130559. PMID 20566619